CLINICAL TRIAL: NCT02629640
Title: Enhanced CJD Surveillance in the Older Population
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Department of Health, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15/SS/0196
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Prion Disease; Dementia
Keywords: vCJD; prion disease; dementia; old-age; surveillance; brain banking; public health
MeSH Terms: conditions — Prion Diseases; Dementia | interventions — Blood Specimen Collection; Autopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples
  * Buccal samples
  * Brain tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Research Participants: Medical history questionnaire; clinical assessment and review; participant follow-up; blood or buccal sample; post mortem examination.
  Interventions: Other: Medical history questionnaire; Other: Clinical assessment and review; Other: Participant follow-up; Other: Blood or buccal sample; Other: Post mortem examination

INTERVENTIONS:
Other: Medical history questionnaire — Epidemiological review of past medical/dental history; residential history; occupational history; family history of neurodegenerative disease.
Other: Clinical assessment and review — History of current illness; neurological examination including general appearance, full cognitive assessment and physical examination; MRI research brain scan.
Other: Participant follow-up — Hospital patient management system; regular telephone contact with patient/representative.
Other: Blood or buccal sample — Codon-129 genotyping; storage for future research.
Other: Post mortem examination — Brain tissue donation to the Edinburgh Brain and Tissue Bank for research,including investigations for evidence of prion disease.

SUMMARY:
The purpose of this study to investigate if cases of Creutzfeldt-Jakob Disease (CJD) and other forms of prion disease are being missed in older adults living within Lothian.

DETAILED DESCRIPTION:
The study involves patients aged 65 years or over who have been seen by a neurologist or psycho-geriatrician and identified as having features that are atypical for the known types of dementia. All patients will be invited to an initial meeting with the research team to discuss the study and, if they agree to participate, for clinical assessment and epidemiological review. Participants will be asked to donate blood or a buccal sample for codon-129 polymorphism genotyping and may be offered a MRI brain scan if no such imaging has been previously undertaken. Participants will also be asked to consider if, in the event of their death, they would donate samples of brain tissue to the Edinburgh Brain Bank for use in this and future research. Telephone follow up will be offered within 1 month of joining the study and at 3 monthly intervals thereafter, with further clinical review offered if deemed appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or above
* Patients accessing NHS Lothian neurology and psychogeriatric services
* Patients who have features atypical for the recognised forms of dementia
* Appropriate informed consent

Exclusion Criteria:

* Patients aged below 65 at time of recruitment
* Patients diagnosed with a clear alternative demonstrable pathology

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65+ accessing NHS Lothian neurology/psychogeriatric services with atypical features of the recognised forms of dementia. Eligible patients will be identified by the local clinical team by screening their existing patient lists, as they see patients as they attend their clinic or are visited in the community. The clinic staff are asked to consult the study team to confirm the patient's eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Evidence of prion disease pathology in the Lothian population, a description of the associated clinical/pathological and epidemiological features and referral characteristics, and how this compares with other cases of prion disease. | 4.5 years

SECONDARY OUTCOMES:
Description of clinical, pathological and epidemiological characteristics of patients with atypical features of dementia in the Lothian population. | 4.5 years
Assessment of the suitability of methods to support an extended system of enhanced CJD surveillance in the rest of the UK. | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Molesworth, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- CJD Research and Surveillance Unit, Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No